CLINICAL TRIAL: NCT01633840
Title: New Validated Recipes for Double-blind Placebo-controlled Low Dose Food Challenges
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Christina West (Other)
Collaborators: The Västerbotten county council (Unknown); State Government founding for Health Care research (Unknown); Oskarsfonden (Unknown); Nutricia, Inc. (Industry)
Responsible Party: Sponsor-Investigator, Christina West, MD, PhD, Umeå University
Organization: Umeå University (Other)
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Diagnostic
Other Study IDs: 06-089M
Record Dates: First submitted 2012-06-20; First posted 2012-07-04 (Estimated); Last update posted 2021-04-30 (Actual); Status verified 2021-04

CONDITIONS: Allergy
Keywords: double-blind placebo-controlled food challenges; food allergy; food hypersensitivity; triangle test; validated recipes
MeSH Terms: conditions — Hypersensitivity; Food Hypersensitivity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Elemental E028 with added food allergens (Active Comparator)
  Interventions: Other: Elemental E028 with added food allergens
- Elemental E028 (Placebo Comparator)
  Interventions: Other: Elemental E028

INTERVENTIONS:
Other: Elemental E028 with added food allergens — Test materials containing liquid vehicle (Elemental E028)with added food allergens (active)
  Arms: Elemental E028 with added food allergens
Other: Elemental E028 — Elemental E028 with no added food allergens
  Arms: Elemental E028

SUMMARY:
This study aimed to validate new recipes for cow's milk, hen's egg, soy, cod and wheat, to be used in blinded low-dose food challenges.

ELIGIBILITY:
Inclusion Criteria:

* Children belonging to one of two age groups: 7-8 years or 14-15 years
* No previous hypersensitivity reaction to the food to be tested
* Capacity to understand the test instructions and to participate in the test sessions

Exclusion Criteria:

* Children not belonging to one of the two age groups: 7-8 years or 14-15 years
* One or more previous hypersensitivity reaction to the food to be tested
* Unability to understand the test instructions and to participate in the test sessions

Ages: 8 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 275 (Actual)
Dates: Start 2008-09; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Number of participants detecting sensorial differences between the active materials (containing the allergens cow's milk, hen's egg, soy, wheat or cod) and the placebo materials
  The present study aimed to validate new recipes for low-dose double-blind placebo-controlled food challenges in school children, by assessing that no sensory differences between the active materials containing cow's milk, hen's egg, soy, wheat or cod, and the placebo materials could be detected by test panels.

CONTACTS AND LOCATIONS:
Overall Officials: Christina E West, MD, PhD, Principal Investigator — Umeå University Sweden
Locations (1):
- Department of Clinical Sciences, pediatrics, Umeå, Sweden

REFERENCES:
- [Background] Winberg A, Nordstrom L, Strinnholm A, Nylander A, Jonsall A, Ronmark E, West CE. New validated recipes for double-blind placebo-controlled low-dose food challenges. Pediatr Allergy Immunol. 2013 May;24(3):282-7. doi: 10.1111/pai.12061. PMID 23590418